CLINICAL TRIAL: NCT02098031
Title: Improving the Nutrition Status of 6 to 8 Months Old Children Through Diet Diversification and Better Dietary Intakes in the Kabale and Kisoro Districts in South-Western Uganda
Brief Title: Improving the Nutrition Status of Infants in South-Western Uganda
Acronym: CHNUDEV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Kyambogo University (Other)
Responsible Party: Principal Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Infant Malnutrition; Nutrition Knowledge; Growth; Cognitive Development
Keywords: Child Nutrition Sciences; Growth and Development; Developing Countries
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- intervention (Experimental): Nutritional intervention (nutrition education)
  Interventions: Other: Improving nutrition knowledge among mothers

INTERVENTIONS:
Other: Improving nutrition knowledge among mothers
  Arms: intervention

SUMMARY:
Undernutrition and growth restriction due to poor diet and inadequate nutrient intake continues to be a global challenge, particularly in the developing countries including Uganda. The etiology of inadequate nutrient supply to infants may relate to lack of resources or knowledge or a combination of both. Poor nutrient intake and impaired growth may affect brain and cognitive development.

This study aims to evaluate nutrient intake, growth and cognitive function among children between 6 and 36 months living in the fertile Kabale and Kisoro region in south-western Uganda. The investigators hypothesize that nutrition education to mothers can bring about improved dietary intake and nutritional status among children aged 6-36 months.

A follow-up study was conducted during the period January - July 2022.

ELIGIBILITY:
Inclusion Criteria:

* A lead caretaker with a 6-8 months infant (child/lead caretaker pair) who will have given consent to participate in the study. If there is more than one child of the age in the household, the younger one will be taken as the index/study child.

Exclusion Criteria:

* Is older than 8 months at baseline
* Congenital malformations or physical handicap that may influence growth or interfere with taking of anthropometric measurements
* Disability that will influence nutrient intake
* Been diagnosed with mental or brain illness as evidenced by mother or health worker.
* If the family that is likely to emigrate during the study period

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in the prevalence of stunting (<-2 SD of the WHO, 2006 growth reference standards) | 6-8, 12-16, 20-24 (main outcome time point), 36 months, 7-10 years
  The investigators will measure the change in stunting between the three indicated time points.

SECONDARY OUTCOMES:
Change in mean weight-for-age z-score | 6-8, 12-16 and 20-24, 36 months, 7-10 years
  The investigators will measure the change in mean weight for age z-score between the three indicated time periods.
Change in mean weight-for-height z-score | 6-8, 12-16, 20-24, 36 months, 7-10 years
  The investigators will measure the change in mean weight for height z-score between the three indicated time periods.
Change in mean Mid Upper Arm Circumference (MUAC) z-score | 6-8, 12-16, 20-24, 36 months, 7-10 years
  The investigators will measure the change in MUAC between the three indicated time periods.
Change in mean diet diversification score (DDS) | 6-8, 12-16, 20-24, 36 months
  The investigators will measure the change in DDS between the three indicated time periods.
Change in Ages and Stages Questionnaire Scores (AQS) | 6-8, 12-16, 20-24, 36 months
  The investigators will measure the change in AQS between the three indicated time periods.
Change in The Kaufman Assessment Battery for Children (2nd ed.; KABC-II) and the Test of Variable of Attention (TOVA) | 7-10 years
  The investigators will measure the change in the scores of these tests at indicated time periods.
Change in Bayley Child Development test 3 ed. | 6-8, 12-16, 20-24, 36 months
  The investigators will measure the change in Bayley Child Development test 3 ed. between the three indicated time periods.
Change in gut microbiota | 20-24, 36 months, 7-10 years
  Fecal samples will be collected and the investigators will measure the change in gut microbiota between the three indicated time periods.
Change in oral microbiota | 36 months, 7-10 years
  Saliva samples will be collected and the investigators will measure the change in oral microbiota at indicated time periods.
Change in Mullens test | 36 months
  The investigators will measure the change in Mullens test between the two groups after 36 months.
Change in Becks Depression Inventory II questionnaire to determine the maternal self-reported depression symptoms | 7-10 years
  The investigators will measure the change in this test between the two groups at indicated time periods
Change in the Center for Epidemiological Studies Depression Scale questionnaires to determine the maternal self-reported depression symptoms | 7-10 years
  The investigators will measure the change in this test between the two groups at indicated time periods
Oral health | 7-10 years
  The investigators will assay caries using photographs

CONTACTS AND LOCATIONS:
Locations (1):
- Kyambogo University, Kampala, Uganda

REFERENCES:
- [Derived] Atukunda P, Ngari M, Chen X, Westerberg AC, Iversen PO, Muhoozi G. Longitudinal assessments of child growth: A six-year follow-up of a cluster-randomized maternal education trial. Clin Nutr. 2021 Sep;40(9):5106-5113. doi: 10.1016/j.clnu.2021.08.007. Epub 2021 Aug 20. PMID 34461584
- [Derived] Kakwangire P, Moss C, Matovu N, Atukunda P, Westerberg AC, Iversen PO, Muhoozi G. The association between dietary diversity and development among children under 24 months in rural Uganda: analysis of a cluster-randomised maternal education trial. Public Health Nutr. 2021 Sep;24(13):4286-4296. doi: 10.1017/S136898002100077X. Epub 2021 Mar 12. PMID 33706831
- [Derived] Atukunda P, Muhoozi GK, Diep LM, Berg JP, Westerberg AC, Iversen PO. The association of urine markers of iodine intake with development and growth among children in rural Uganda: a secondary analysis of a randomised education trial. Public Health Nutr. 2021 Aug;24(12):3730-3739. doi: 10.1017/S1368980020001603. Epub 2020 Jul 13. PMID 32654677
- [Derived] Atukunda P, Muhoozi GKM, van den Broek TJ, Kort R, Diep LM, Kaaya AN, Iversen PO, Westerberg AC. Child development, growth and microbiota: follow-up of a randomized education trial in Uganda. J Glob Health. 2019 Jun;9(1):010431. doi: 10.7189/jogh.09.010431. PMID 31131103
- [Derived] Muhoozi GKM, Atukunda P, Diep LM, Mwadime R, Kaaya AN, Skaare AB, Willumsen T, Westerberg AC, Iversen PO. Nutrition, hygiene, and stimulation education to improve growth, cognitive, language, and motor development among infants in Uganda: A cluster-randomized trial. Matern Child Nutr. 2018 Apr;14(2):e12527. doi: 10.1111/mcn.12527. Epub 2017 Sep 19. PMID 28925580